CLINICAL TRIAL: NCT00233636
Title: A 2 Part Phase 2 Trial to Evaluate ZD1839 (Iressa™) & Radiotherapy in Patients w/Locally Advanced Inoperable Squamous Cell Carcinoma of the Head & Neck
Brief Title: Iressa and Radiotherapy in the Treatment of the Locally Advanced Inoperable Squamous Cell Carcinoma of the Head and Neck
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1839IL/0070
Record Dates: First submitted 2005-10-04; First posted 2005-10-06 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2011-01

CONDITIONS: Head and Neck Cancer; Carcinoma, Squamous Cell
Keywords: Squamous Cell Carcinoma of Head and Neck; Inoperable locally advanced Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck | interventions — Gefitinib; Radiotherapy

INTERVENTIONS:
Drug: Iressa (Gefitinib)
Procedure: Radiotherapy

SUMMARY:
The aim of the study is to determine if Iressa added to radiotherapy is effective and safe in shrinking tumour dimensions.

ELIGIBILITY:
Inclusion Criteria:

* Histologically Confirmed locally advanced Squamous Cell Carcinoma of Head and neck
* At least one measurable tumour lesion

Exclusion Criteria:

* No previous treatment such as chemotherapy, radiotherapy and/or surgery for Carcinoma Head and Neck
* No other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ
* Any evidence of severe or uncontrolled systemic disease (e.g. unstable or uncompensated respiratory, cardiac, hepatic or renal disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28
Dates: Start 2003-07

PRIMARY OUTCOMES:
Tumour Response Rate, as complete response (CR) and partial response (PR) . Six months after Last Patient In.

SECONDARY OUTCOMES:
Time to progression, Overall survival, Duration of response. Six months after Last Patient In.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Italy Medical Director, MD, Study Director — AstraZeneca
Locations (6):
- Italy (6):
  - Research Site, Aviano
  - Research Site, Azienda
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Palermo
  - Research Site, Ragusa